CLINICAL TRIAL: NCT00539383
Title: A Phase 1, Open-Label, Dose Escalation Study of ANG1005 in Patients With Advanced Solid Tumors and Metastatic Brain Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Angiochem Inc (Industry)
Responsible Party: Jean-Paul Castaigne, MD - President & CEO, Angiochem Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ANG1005-CLN-02; FDA
Record Dates: First submitted 2007-10-03; First posted 2007-10-04 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Advanced Solid Tumors With and Without Brain Metastases
Keywords: Lung cancer; Breast cancer; Melanoma; Hepatocellular carcinoma; Brain metastases
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Melanoma; Carcinoma, Hepatocellular; Brain Neoplasms | interventions — paclitaxel-Angiopep-2 conjugate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: ANG1005

INTERVENTIONS:
Drug: ANG1005 — IV infusion once every 21 days

SUMMARY:
This is a phase 1, multi-centre, sequential cohort, open-label, dose-escalation study of the safety, tolerability, and PK of ANG1005 in patients with solid tumors (with or without brain metastases). ANG1005 will be given by IV infusion once every 21 days (1 treatment cycle). Each patient will participate in only 1 dose group and will receive up to 6 cycles of treatment provided there is no evidence of tumor progression, there is recovery to ≤Grade 1 or baseline nonhematologic, ANG1005-related toxicity (except alopecia), the absolute neutrophil count is ≥1.5 x 109/L, and the platelet count is ≥100 x 109/L.

DETAILED DESCRIPTION:
This is a phase 1, multi-centre, sequential cohort, open-label, dose-escalation study of the safety, tolerability, and PK of ANG1005 in patients with solid tumors (with or without brain metastases). ANG1005 will be given by IV infusion once every 21 days (1 treatment cycle). Each patient will participate in only 1 dose group and will receive up to 6 cycles. Patients may receive additional cycles of ANG1005 if there is no evidence of tumor progression, there is recovery to ≤Grade 1 or baseline nonhematologic, ANG1005-related toxicity (except alopecia), the absolute neutrophil count is ≥1.5 x 109/L, and the platelet count is ≥100 x 109/L.

Initially, cohorts of 1 - 3 patients will be enrolled into each dose group. Dose escalation by dose doubling will be done for the first 3 dose groups followed by a modified Fibonacci dose escalation scheme with increases of 67%, 50%, 40% and 33% thereafter. If 1 or more patients in a cohort experience an emergent ≥ Grade 2 drug-related toxicity during the first treatment cycle, then a minimum of 3 patients will be enrolled into that, and all subsequent cohort(s) and dose doubling will be stopped if applicable.

If > 1 patient in a cohort experience a dose limiting toxicity (DLT) during the first treatment cycle, defined as any of the following that are both treatment-emergent and at least possibly related to ANG1005: i) Any Grade 3 or 4 nonhematologic toxicity, ii) Febrile neutropenia, iii) Grade 4 neutropenia of ≥7 days duration, and/or iv) Any Grade 4 thrombocytopenia, then dose escalation will stop and prior doses will be explored as the maximum tolerated dose (MTD), that dose-level at which ≤1 of 6 patients in a cohort develop an emergent DLT).

Once the MTD is established, approximately 14 patients will be enrolled at that dose-level in order to further assess the safety and tolerability of ANG1005, the PK profile of ANG1005 at the MTD, and the preliminary anti-tumor activity of ANG1005 in patients with solid tumors (with or without brain metastases).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Histologically or cytologically confirmed metastatic or advance-stage solid tumor that has progressed following standard therapy or for which, in the opinion of the Investigator, no standard effective therapy is available; patients without brain metastases may be enrolled into the dose-escalation part of the study
3. Patients enrolled into the expanded MTD cohort must have shown unequivocal evidence of brain metastases
4. Male and female patients.
5. Age ≥18 years
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
7. An expected survival of at least 3 months
8. Measurable disease according to RECIST criteria; patients with brain metastases must have at least one measurable lesion in the brain, according to RECIST criteria
9. Male and female subjects who are not surgically sterile or post-menopausal must agree to use reliable methods of birth control for the duration of the study and for 90 days after the last dose of study drug administration; male partners of female subjects should use condoms for the duration of the study, and for 90 days after the last dose of study drug administration

Exclusion Criteria:

1. Chemotherapy, radiotherapy (except palliative radiation delivered to <20% of bone marrow), or investigational agents within 4 weeks before the first dose of study drug. Biologic therapy (such as 13-cis-retinoic acid, thalidomide, tamoxifen, celebrex, erlotinib, imatinib, vorinostat, and lapatinib) and immunotherapy (such as interferon a or b, cdx-110 (EGFR vIII vaccine), interleukin 2, thalidomide) within 1 week before the first dose of study drug. Bevacizumab within 6 weeks before the first dose of study drug
2. Pregnant or lactating females
3. Any acute viral, bacterial, or fungal infection that requires parenteral therapy within 14 days prior to study treatment
4. Known severe hypersensitivity to paclitaxel
5. Severe toxicity with previous taxane treatment
6. Treatment with P450 CYP 3A4 or CYP 2C8 enzyme-inducing anti-convulsant drugs within 14 days prior to treatment with study drug
7. Patients with inadequate hematological, liver, and renal function
8. Known or suspected acute or chronic active Hepatitis B, Hepatitis C, or HIV/AIDS
9. Patients with unstable or uncompensated respiratory, cardiac, hepatic or renal disease or any other organ system dysfunction, medical condition, or laboratory abnormality which, in the opinion of the Investigator, would either comprise the patient's safety or interfere with the evaluation of the test material
10. Evidence of persistent Grade 2 or greater neurotoxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To characterize the safety and tolerability of intravenously administered ANG1005 in patients with advanced solid tumors and metastatic brain cancer. | On-going
To identify the maximum tolerated dose (MTD) of ANG1005 in patients with advanced solid tumors and metastatic brain cancer. | End of dose escalation

SECONDARY OUTCOMES:
To examine the pharmacokinetics (PK) of ANG1005. | End of study
To confirm the safety and tolerability of ANG1005 at the MTD. | End of dose escalation
To assess the immunogenicity of ANG1005. | End of study
To obtain preliminary information on the antitumor activity of ANG1005 in patients with advanced solid tumors with brain metastases. | On-going

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Gabrail Cancer Center, Canton, Ohio
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
  - UT Health Science Center, Cancer Therapy and Research Center, San Antonio, Texas

REFERENCES:
- [Result] Kurzrock R, Gabrail N, Chandhasin C, Moulder S, Smith C, Brenner A, Sankhala K, Mita A, Elian K, Bouchard D, Sarantopoulos J. Safety, pharmacokinetics, and activity of GRN1005, a novel conjugate of angiopep-2, a peptide facilitating brain penetration, and paclitaxel, in patients with advanced solid tumors. Mol Cancer Ther. 2012 Feb;11(2):308-16. doi: 10.1158/1535-7163.MCT-11-0566. Epub 2011 Dec 27. PMID 22203732
- See also: Related Info — http://www.angiochem.com